CLINICAL TRIAL: NCT04741126
Title: Effectiveness of the Manually Assisted Cough Technique on Peak Coughs Flow and Pulmonary Functions in Patients With Incomplete Cervical Spine Injury
Brief Title: Manually Assisted Cough Technique and Incomplete Cervical Spine Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rec/00782 Nadeem Ahmad
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Spinal Cord Injuries
Keywords: Manually assisted cough technique; Peak cough flow; Pulmonary function; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Protocol (Experimental): Hospital-based manually assisted cough technique for 4 weeks.
  Interventions: Other: Manually assisted cough technique

INTERVENTIONS:
Other: Manually assisted cough technique — Manually assisted cough technique will be given for four weeks. 10 to 12 repetitions of manually assisted cough technique with rest will be given in one minute 3 to 4 time of repetition in a 1 set. The result of the peak cough flow meter and incentive spirometer will be check pre and post only.3 sets will be given in one session and 2-time session will be recommended per day. The session will be given three days in a week. The Result of the Peak Cough flow meter and incentive spirometer will be check pre and post only.

SUMMARY:
To determine the effectiveness of manually assisted cough technique on peak cough flow and pulmonary functions in patients with incomplete cervical spine injury. Previous studies were designed to target only a small sample. Level and American Spinal Cord Injury Association (ASIA) scale were not specified so this study covers this aspect.

DETAILED DESCRIPTION:
The previous studies show that the partial control of the muscle necessary for cough, which varies with motor level, proportionately improves the patient's ability to cough volitionally. Spinal cord injury also affects mucus clearance, the peak flow meter was used to assist the ability of cough and they also measure the peak cough flow (PFC).In the literature for the airway clearance, the following techniques were used, incentive spirometer, balloon, and blowing exercise, manually assisted cough technique active cycle of breathing exercise, postural drainage, autogenic drainage, positive expiratory pressure. There is increasing interest in strategies such as interval training that may provide a tolerable training load while maintaining an effective stimulus for adaptation. Manually assisted cough technique is used to enhance the cough strength, to help with mucus secretion it can be carried out in lying, side-lying, or sitting positions.it is important that clear secretion in order to maintain clear and healthy lungs, the risk of repeated chest infection and complication can be reduced which improve the quality of life. Manually assisted cough is a technique using strong arms to assist cough. This may be providing help in neuromuscular disease or spinal cord injury with weak respiratory and abdominal muscle.

ELIGIBILITY:
Inclusion Criteria:

* The patient with incomplete cervical spine injury at C4, C5,
* bronchitis,
* shortness of breath having Peak cough flow (PCF) less than 50% and
* ASIA impairment scale C &D

Exclusion Criteria:

* The patient with upper cervical,
* thoracic, and
* lumbar spine injury,
* diagnosed with TB,
* degenerative diseases,
* surgical conditions, and
* complete spinal cord injury.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Peak cough flow | 4 weeks
  Changes from the baseline will be measured after 4 weeks through a small, hand-held device which is used to monitor a person's ability to breathe out air. It measures the airflow through the bronchi of the lungs and thus indicates the degree of obstruction in the airways. Peak flow readings are higher health airways and decreases in obstructive airways.

SECONDARY OUTCOMES:
Pulmonary functions | 4 weeks
  Changes from the baseline will be measured after 4 weeks through the incentive spirometer. This device will measure how deeply patient can inhale (breathe in) and to evaluate the volumes and capacities of the patient before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mehwish Waseem, MSPT(CPPT), Principal Investigator — Riphah International University
Locations (1):
- Paraplegic center Peshawar., Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parmar K, Gunjal SB. Effectiveness of Manually Assisted Cough Technique on Peak Cough Flow in Patients with Spinal Cord Injury. Int J Res Rev. 2020;7(2):243-8.
- [Background] Choi WA, Park JH, Kim DH, Kang SW. Cough assistance device for patients with glottis dysfunction and/or tracheostomy. J Rehabil Med. 2012 Apr;44(4):351-4. doi: 10.2340/16501977-0948. PMID 22453774
- [Background] Beauchamp MK, Nonoyama M, Goldstein RS, Hill K, Dolmage TE, Mathur S, Brooks D. Interval versus continuous training in individuals with chronic obstructive pulmonary disease--a systematic review. Thorax. 2010 Feb;65(2):157-64. doi: 10.1136/thx.2009.123000. Epub 2009 Dec 8. PMID 19996334
- [Background] Brown R, DiMarco AF, Hoit JD, Garshick E. Respiratory dysfunction and management in spinal cord injury. Respir Care. 2006 Aug;51(8):853-68;discussion 869-70. PMID 16867197